CLINICAL TRIAL: NCT04486235
Title: A Randomized, Controlled Pilot Study of a Patient-Initiated Approach to Increasing Weight Communication in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1812006829
Record Dates: First submitted 2019-04-25; First posted 2020-07-24 (Actual); Results first posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2020-04

CONDITIONS: Obesity; Primary Care; Health Communication
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Randomization is stratified. On the screening form, participants indicate whether or not they plan to speak with their physician about their weight in their appointment. Randomization is stratified by if if the participant indicates that they plan to speak about weight or not.
Masking Description: The condition of the participant is revealed after the participant completes the consent form and screening questionnaire and is deemed eligible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receive experiential pamphlet
  Interventions: Behavioral: Brief waiting room pamphlet
- Control (No Intervention): No materials, usual care

INTERVENTIONS:
Behavioral: Brief waiting room pamphlet — An experiential pamphlet including brief assessment questions and recommended questions for the participant to ask their physician based on their responses. Areas covered in the pamphlet include patients' knowledge of weight status and implications of weight, confidence in physicians' abilities to treat weight, stage of change for weight-related behaviors, and comfort in discussing their weight.
  Arms: Intervention

SUMMARY:
This study tests the feasibility, acceptability, and preliminary efficacy of using a brief pamphlet in the primary care waiting room focused on promoting patient-initiated weight-related discussions in primary care appointments.

DETAILED DESCRIPTION:
Obesity is a chronic and complex disease that many national and professional organizations recommend be discussed frequently in primary care. However, rates of weight-related communication in primary care are suboptimal. When patients and physicians communicate about weight (defined as usage of any the 5As-ask, assess, advise, agree, and/or assist-in a weight-related conversation), patients are more likely to improve dietary habits, demonstrate more motivation for health behavior change, attempt weight loss treatment, and lose more weight as compared to patients who do not engage in weight-related communication with their physicians. Interventions have attempted to increase the rates of weight-related communication in primary care. However, they have focused solely on physicians and have only yielded modest efficacy. Intervention with patients on proposed patient-related barriers may be key to improving the rate of weight-related communication in primary care. The waiting room prior to appointments is an underutilized intervention setting. Prior waiting room interventions have shown promising results for increasing health communication between patients and physicians. However, no prior study has focused on weight-related communication. Thus, this study aims to test the feasibility, acceptability, and preliminary efficacy of an experiential pamphlet delivered in the waiting room targeting patient-related barriers to weight communication.

ELIGIBILITY:
Inclusion Criteria:

* Present for an appointment at the Family Medicine Office
* Indicate that they can speak and read English
* Indicate that their Shape is > or = 5 on measure (Stunkard, Sørensen, & Schulsinger, 1983)
* Indicate that they are 18 years or older

Exclusion Criteria:

- Indicate that they are Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Remmert, MS, Principal Investigator — Drexel University
Locations (1):
- Drexel University Family Medicine Office, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 32 | 30
Analysis | 30 | 30
Completed | 30 | 30
Not Completed | 2 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (15.4) | 38.2 (16.02) | 40.6 (15.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 17 | 14 | 31
  Female | 13 | 15 | 28
  Transgender | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 29 | 29 | 58
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 10 | 21
  White | 16 | 15 | 31
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Treatment Acceptability Questionnaire
Description: Intervention participants reported acceptability, as measured by the Treatment Acceptability Questionnaire (Hunsley, 1992). This is a 6-item scale that asks the participant to rate several metrics of acceptability with Likert scale responses (individual items range 1-7, one item is reverse scored). A higher score indicates greater acceptability, a score of 21 is the benchmark for acceptability. Overall range of 6-42.
Time Frame: Immediately after appointment (Same day as intervention delivery)
Population: Only intervention participants saw the pamphlet and provided acceptability feedback
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 0
units on a scale | 35.8 (5.5) |

2. Primary Outcome: Feasibility of Recruitment From Primary Care Waiting Room and Intervention Delivery
Description: Study flow will be tracked by study staff and compared to pre-determined benchmarks. 1) Percentage of patients who indicate verbal consent for screening (benchmark >70%), 2) percentage of eligible participants after screening (benchmark >50%), 3) percentage of participants who refuse to participate because of focus on weight (benchmark <20%), 4)percentage of participants who complete the experiential pamphlet (benchmark >80%).
Time Frame: When study staff is recruiting in the office during the data collection period, approx. 20 days over 6 months
Population: Tracked by participant flow, 295 participants invited to participate by research staff, eventually resulting 135 assessed for eligibility, and ultimately 62 randomized
Measure: Number; unit: percentage of participants
Groups:
- Feasibility, Tracked by Participant Flow: Feasibility was measured by tracking flow and calculating: 1) Percentage of patients who indicate verbal consent for screening, 2) percentage of eligible participants after screening, 2) percentage of participants who refuse to participate because of focus on weight, 3)percentage of participants who complete the experiential pamphlet. Study flow will be tracked by study staff and compared to pre-determined benchmarks
Arm/Group | Feasibility, Tracked by Participant Flow
Number analyzed (Participants) | 295
percentage of participants
  Percentage of participants indicated verbal consent for screening | 60
  Percentage of eligible participants after screening: number analyzed (Participants) | 115
  Percentage of eligible participants after screening | 53.5
  Percentage of screened participants who refuse to participate because of focus on weight: number analyzed (Participants) | 115
  Percentage of screened participants who refuse to participate because of focus on weight | 0
  Percentage of participants who complete the experiential pamphlet: number analyzed (Participants) | 30
  Percentage of participants who complete the experiential pamphlet | 86.2

3. Secondary Outcome: If Weight Was Spoken About in the Appointment
Description: Participants respond to Yes/No questions about content of their appointment
Time Frame: Immediately after appointment (Same day as intervention delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 30
Participants
  Patient-initiated weight discussion occured | 7 | 5
  Patient- or physician-initiated weight discussion occurred | 14 | 11

ADVERSE EVENTS:
Time Frame: Collected data from participants during primary care appointment (approx. 15-90 min), data collection occurred over a period of 6 months
Description: This was a brief, low risk study of providing a pamphlet about health and weight to patients in the waiting room before a primary care appointment
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/30
Other Adverse Events (participants affected / at risk) | 0/32 | 0/30

LIMITATIONS AND CAVEATS:
Small sample size, location for study was primarily staffed by Family Medicine residents which may limit generalizability

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT04486235/Prot_SAP_000.pdf